CLINICAL TRIAL: NCT04054063
Title: An Open Label, Single-Center, Single Dose Combination of HSK3486 and Etomidate Intravenous Bolus Injection to Determine the Safety, Pharmacodynamics and Pharmacokinetics for Induction of Anesthesia in Healthy Male Subjects
Brief Title: A Study Evaluating Safety, Pharmacodynamics and Pharmacokinetics of HSK3486 and Etomidate for Induction of Anesthesia in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-Australian-04
Record Dates: First submitted 2019-07-04; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2017-06

CONDITIONS: General Anesthetic; Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK3486+etomidate (Experimental): Cohort 1: HSK3486 0.324 mg/kg + etomidate 0.15 mg/kg Cohort 2: HSK3486 0.216 mg/kg + etomidate 0.2 mg/kg Cohort 3: HSK3486 0.432 mg/kg + etomidate 0.1 mg/kg There were an additional 2 cohorts (Cohorts 4 and 5) planned for dose escalation once the optimal ratio of the drug combination was identified from the first 3 cohorts. However, these 2 cohorts were not done as the results of Cohorts 1 to 3 suggested that dose increases would cause higher occurrence of drug-related adverse events (AEs).
  Interventions: Drug: HSK3486+ etomidate

INTERVENTIONS:
Drug: HSK3486+ etomidate

SUMMARY:
This study is designed as an open label, single dose combination of HSK3486 and etomidate in healthy adult male subjects. The study will evaluate the anesthetic/sedation effect of the combination of the 2 drugs and the safety profile including pain on injection, hypotension, tachycardia or bradycardia effects (HSK3486), and involuntary muscle movements, nausea and vomiting potential and adrenal suppression (etomidate).

All subjects will be administered HSK3486 plus etomidate. Subjects will be confined to the study unit from the evening of Day -1 until the morning of Day 2, then will be required to return for a follow up visit on Day 7.

Intensive PD, PK, safety and tolerability and assessments will be performed prior to dosing on Day 1 until 24 hours post-dose (Day 2).

ELIGIBILITY:
Inclusion Criteria:

* 1.Male, aged 18 - 49 years (inclusive)
* 2.Be in general good health without clinically significant medical history, as determined by the investigator
* 3.American Society of Anesthesiologists Physical Status Classification of I or II
* 4.Body mass index (BMI) between 18 and 30 kg/m2 (inclusive)
* 5.Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen, hepatitis C and Human Immunodeficiency Virus (HIV) at screening; and drugs of abuse, alcohol pre dose on Day -1
* 6.Normal or non-clinically significant findings on a physical examination, 12-lead ECG and vital signs (respiration rate between 12 and 20 breaths per minute, BP between 100-140/50-90 mmHg, heart rate between 45-99 beats per minute, temperature between 35.8 degrees and 37.5 degrees). Pulse oximetry values >95% on room air.
* 7.Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the investigator decides that out-of-range values are not clinically significant
* 8.Ability to provide written informed consent
* 9.Willing and able to follow study instructions and likely to complete all study requirements
* 10.Suitable venous and arterial access.

Exclusion Criteria:

* 1.History of allergy or sensitivity to: propofol, etomidate or components of HSK3486 (excipients soy bean oil, glycerine, triglycerides, purified egg phospholipids, sodium oleate and sodium hydroxide), or plain lignocaine
* 2.History of clinically significant problems with anesthesia induction
* 3.Current smoker, or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within 2 months prior to screening
* 4.History of excessive alcohol intake (more than 4 standard drinks daily, on average) or use of recreational drugs within the last 3 months prior to screening
* 5.Intake of > 8 caffeine-containing drinks per day, on average, or approximately 800mg of caffenine daily on average; history of intolerance of abstinencce from caffeine for 3 days
* 6.Use of prescription or over the counter medications within 7 days of investigational product administration, with the exception of paracetamol, oral non-steroidal anti-inflammatory agents, topical over the counter preparations and routine vitamins (if they do not exceed the recommended daily dose), unless agreed as non-clinically relevant by the investigator and sponsor.
* 7.Standard donation of blood within 30 days of the study
* 8.Donation of plasma or participation in a plasmapheresis program within 7 days of investigational product administration
* 9.Receipt of any investigational study drug within 30 days prior to screening
* 10.Unable to fast for the 6 hours prior to investigational product administration
* 11.Clinically significant (as judged by the investigator) presence of acute illness (e.g. gastrointestinal illness, infection such as influenza, upper respiratory tract infection) at admission to the clinical study unit
* 12.Anticipated need for surgery or hospitalization during the study
* 13.Craniofacial abnormality that would potentially interfere with airway management under unconscious sedation or anesthesia
* 14.History of seizures or epilepsy
* 15.History of ischaemic heart disease
* 16.History of brady- or tachy-dysrhythmias requiring medical care
* 17.History of asthma, with bronchospasm requiring treatment in the last 3 months
* 18.Any condition, which in the investigator's opinion, puts the subject at significant risk, could confound the study results or may interfere significantly with the subject's participation in the study
* 19.Receipt of HSK3486 less than 4 weeks prior to the start of the study.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Safety by measurement of Adverse Events | on day 1 until 24 hours post-dose

SECONDARY OUTCOMES:
Richmond Agitation Sedation Scale (RASS) | First dose of study drug on day 1
  * 0 Alert and calm
  * 1 Not fully alert, but has sustained awakening (eyeopening/eye contact) to voice (≥ 10 seconds)
  * 2 Briefly awakens with contact to voice (< 10 seconds)
  * 3 Movement or eye opening to voice (but no eye contact)
  * 4 No response to voice, but movement or eye opening to physical stimulation
  * 5 No response to voice or physical stimulation
bispectral index (BIS) | First dose of study drug on day 1
subject-rated Quality of Recovery Assessment (QoR-9） | First dose of study drug on day 1
Peak concentration (Cmax) | on day 1 until 24 hours post-dose
Time to plasma peak concentration(Tmax) | on day 1 until 24 hours post-dose
Area Under the Curve | on day 1 until 24 hours post-dose